CLINICAL TRIAL: NCT05233579
Title: Open-Label Trial of Sulforaphane in Premutation Carriers With FXTAS to Find Biomarkers
Brief Title: Open-Label Trial of Sulforaphane in Premutation Carriers With FXTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 1743661
Record Dates: First submitted 2021-10-20; First posted 2022-02-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Fragile X Associated Tremor/Ataxia Syndrome (Fxtas) (Diagnosis)
Keywords: Sulforaphane
MeSH Terms: conditions — Fragile X Tremor Ataxia Syndrome; Disease | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sulforaphane 1 Tablet (Experimental): Participants are taking 1 tablet per day. All participants will start with 1 tablet and continue with 1 tablet for 2 weeks before increasing dose.
  Interventions: Dietary Supplement: Sulforaphane
- Sulforaphane 2 Tablets (Experimental): Participants will increase dosage to 2 tablets per day after 2 weeks from the start of study participation. Participants will continue to take 2 tablets for 2 addiitonal weeks before increasing dose. If participants experience adverse side effects, participants will decrease dosage to 1 tablet.
  Interventions: Dietary Supplement: Sulforaphane
- Sulforaphane 3 Tablets (Experimental): Participants will increase dosage to 3 tablets per day at 4 weeks from the start of study participation. Participants will continue to take 3 tablets for 2 addiitonal weeks before increasing dose. If participants experience adverse side effects, participants will decrease dosage to 2 tablets.
  Interventions: Dietary Supplement: Sulforaphane
- Sulforaphane 4 Tablets (Experimental): Participants will increase dosage to 4 tablets per day at 6 weeks from the start of study participation. Participants will continue to take 4 tablets for 2 addiitonal weeks before increasing dose. If participants experience adverse side effects, participants will decrease dosage to 3 tablets.
  Interventions: Dietary Supplement: Sulforaphane
- Sulforaphane 5 Tablets (Experimental): Participants will increase dosage to 5 tablets per day at 8 weeks from the start of study participation. Participants will continue to take 5 tablets for 2 addiitonal weeks before increasing dose. If participants experience adverse side effects, participants will decrease dosage to 4 tablets.
  Interventions: Dietary Supplement: Sulforaphane
- Sulforaphane (Experimental): Participants will increase dosage to 6 tablets per day at 10 weeks from the start of study participation. Participants will continue to take 6 tablets for 2 addiitonal weeks before increasing dose. If participants experience adverse side effects, participants will decrease dosage to 5 tablets.
  Interventions: Dietary Supplement: Sulforaphane

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Sulforaphane will be taken one tablet in the morning with breakfast and then every 2 weeks, the dose will be increased by one tablet until a total of 6 tablets are taken in the morning. The supplement should be taken around the same time each day.
  Other Names: Avmacol

SUMMARY:
FXTAS is a rare genetic progressive neurodegenerative disorder, linked to a trinucleotide repeat expansion in the FMR1 gene. FXTAS is characterized by tremor and ataxia in addition to atrophy and white matter disease in the central nervous system (CNS). In addition to the major clinical observations of intention tremor and gait dysfunction, minor symptoms of parkinsonism, neuropathy, and cognitive decline also significantly impact individuals with FXTAS.

The dietary supplement being tested in this study is called Sulforaphane. It is found in broccoli and similar cruciferous vegetables and may cause some gas and discomfort. This is not a study looking at clinical efficacy but instead a study of molecular outcome measures. Investigators want to get more information about how Sulforaphane affects specific biomolecular markers captured in blood.

In this study, participants will be taking an increasing amount of the Sulphoraphane supplement pills (238mg/tablet), starting at 1 and increasing to 6, every morning at breakfast for 6 months. In addition, there will be a total of 3 visits (Initial, 3-month and 6-month) to the MIND Institute where participants will be evaluated. At each visit (3 total) participants will undergo a battery of medical and neurologic exams which make take 2-3 days to complete each time. Participants and/or their caregivers will also be asked to fill out questionnaires/surveys. At the initial visit and at 6 months, we will collect blood for analysis. Two MRI scans will be done, also at the initial visit and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FXTAS
* Presence of a FMR1 premutation (55 to 200 CGG repeats)

Exclusion Criteria:

* Individuals with severe renal failure (GFR is <60 ml/min/1.73 m^2)
* Significant and current reported substance abuse
* Individuals with substance use disorder (meets 6 or more symptoms of substance use disorder criteria)
* Any subject on hospice or on home oxygen
* Individuals who are pregnant

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in mitochondrial function via mitochondrial membrane potential and mass. | Baseline, 6 months
  Primary measures are performed on PBMCs. Mitochondrial mass and membrane potential will use selected floors and either plate readers or analytical flow cytometry.
Changes in mitochondrial function via ATP production | Baseline, 6 months
  Using PMBCs we will observe in changes in ATP production of various segments of the electron transport chain by utilizing different substrates and coupling between electron transport and ATP production.
Observing changes in candidate molecular biomarkers in FXTAS and mitochondrial dysregulation: GRP78 | Baseline, 6 months
  Observing levels in potential molecular biomarkers that affect mitochondrial dysregulation. GRP78 is a master controller of the mitochondrial ER stress response. It helps improve Ca2+ transfer and mitochondrial function. Its level will be measured via ELISA
Observing changes in candidate molecular biomarkers in FXTAS and mitochondrial dysregulation: CHOP level | baseline, 6 months
  Observing levels in potential molecular biomarkers that affect mitochondrial dysregulation. CHOP is a common downstream indicator of mitochondrial ER stress signals. It helps improve Ca2+ transfer and mitochondrial function. Its level will be measured via ELISA
Observing changes in candidate molecular biomarkers in FXTAS and mitochondrial dysregulation: Bax/Bcl-2 ratio | baseline, 6 months
  Observing levels in potential molecular biomarkers that affect mitochondrial dysregulation. Bax/Bcl-2 is a common measure of mitochondrial dysfunction. It helps improve Ca2+ transfer and mitochondrial function. It will be measure via Elisa.

SECONDARY OUTCOMES:
Changes in clinical staging of FXTAS | Baseline, 6 months
  The standardized neurological examination including frontal release signs, snout, jaw jerk, and palmomental reflex; sensory examination of pinprick and vibration sense; and assessment of alternating movements and cranial nerves. These measures constitute the FXTAS Rating Scale (FXTAS-RS).
Changes in subcortical brain structures damaged in FXTAS through MRI imaging | Baseline, 6 months
  The measurements will include anatomic volume for quantifying atrophy. We have developed a robust and efficient method for accurate segmentation of the cerebellum and brainstem and have applied this method to segment the hippocampus, amygdala, basal ganglia, and corpus callosum accurately. We will continue using this method for quantifying volumes of the white matter in individual lobes and subcortical structures, including the corpus callosum, midbrain, pons, and cerebellar white matter, and calibrating iron depositions in subcortical nuclei (i.e., dentate nucleus, substantia nigra, putamen, and globus pallidus)
Changes in FLAIR hypersensitivity volume for subcortical lesions | Baseline, 6 months
  The measurements will include FLAIR hyperintensity volume for subcortical lesions. Subcortical hyperintensities will be segmented automatically using Lesion Prediction Algorithm (LPA) from SPM12, which also co-registers FLAIR images to T1 images. To calculate regional FLAIR hyperintensity volume, we will threshold the generated lesion probability maps at 0.7 and superimpose subcortical and white matter masks to the probability maps using fslmaths from FSL.
Changes in Neurological Quality of Life using the Neuro-QoL upper extremity function fine motor scale | Baseline, 6 months
  The upper extremity function fine motor scale measures the neurological quality of life related to one's ability to carry out various activities involving digital, manual, and reach-related functions ranging from fine motor to self-care. The assessment is administered as a self-report questionnaire and responses are recorded on a scale of 1 (unable to do) to 5 (without any difficulty). The assessment will be administered at baseline and at 6 months and any changes in scaled responses will measure changes in neurological quality of life related to the upper extremity functioning.
Changes in Neurological Quality of Life using the Neuro-QoL lower extremity functioning mobility scale | Baseline, 6 months
  The lower extremity function mobility scale measures the neurological quality of life related to one's ability to carry out various activities involving the trunk region and increasing degrees of bodily movement, ambulation, balance, and endurance. The assessment is administered as a self-report questionnaire and response are recorded on a scale of 1 (unable to do/can't do) to 5 (without any difficulty/no difficulty). The assessment will be administered at baseline and 6 months and any changes in scaled responses will measure change in neurological quality of life related to the lower extremity functioning.
Changes in psychological Issues | Baseline, 6 months
  The Symptom Checklist-90-Revised (SCL-90-R) is a 90 item self-report psychometric questionnaire created to capture a broad range of psychological problems and has been shown to be sensitive in capturing emotional issues in carriers both with and without FXTAS.
Changes in Grip Strength | Baseline, 6 months
  For the NIH Toolbox Grip Strength Test, participants squeeze the Jamar Plus Digital dynamometer as hard as they can for a count of three. The dynamometer provides a digital reading of force in pounds.
Changes in gait variability | Baseline, 6 months
  Gait variability will be measured using the GAITRite in which participants will traverse the GAITRite walkway across 6 walking trials for each condition with minimal interruption.
Changes in dexterity, tremor, and bradykinesia abnormalities | Baseline, 6 months
  The Purdue Pegboard test will measure abnormalities in dexterity, tremor, and bradykinesia.
Changes in kinetic, postural, and rest tremor upper extremity bradykinesia, hypokinesia, dysrhythmia, and dyskinesias | Baseline, 6 months
  Participants will perform pre-defined tasks for the Kinesia One test (e.g., finger to nose, finger tapping, wrist rotation, holding arms extended, arms resting on the legs, and hand grasps).
Changes in cognitive dysfunction using MoCA | Baseline, 6 months
  The Montreal Cognitive Assessment (MoCA) will be administered at baseline and 6 months and the MoCA is scored on a scale of 0-30 points. Changes in the participant's score from the MoCA administered at baseline and the MoCA administered at 6 months will measure whether there are changes in cognitive dysfunction.
Changes in cognitive dysfunction using MMSE | Baseline, 6 months
  The Mini Mental State Exam (MMSE) will be administered at baseline and 6 months. MMSE is scored on a scale of 0-30 points. Changes in participant's score from MMSE administered at baseline and MMSE administered at 6 months will measure whether there are changes in mild cognitive dysfunction.
Changes in executive function deficits using BDS-2 | Baseline, 6 months
  The Behavioral Dysfunction Scale 2 (BDS-2) is a 9-item assessment of simple motor tasks that scores the participant's completion of each item/task on a scale of 0 (patient demonstrates a complete lack of insight into the accuracy of his or her performance and fails to recognize that errors are being made) to 3 (patient demonstrates good performance with no errors). The BDS-2 is administered at baseline and 6 months and changes in participant scores will measure changes in executive function deficits.
Changes in executive function deficits using COWAT | Baseline, 6 months
  The Controlled Oral Word Association Test (COWAT) measures executive functioning deficits using verbal fluency and word retrieval tasks. One's score is calculated by the total number of words listed (1 word = 1 point) Changes in the participant's score from the COWAT administered at baseline and the COWAT administered at 6 months will measure changes in executive function deficits.
Changes in frontal executive planning | Baseline, 6 months
  The Stocking of Cambridge subtest from the CANTAB assessment will be administered to measure deficits in frontal executive planning.
Changes in Hippocampus-mediated memory deficits | Baseline, 6 months
  The Spatial Working Memory and Paired Associates Learning subtest from the CANTAB assessment will be used to measure hippocampus-mediated memory deficits
Changes in motor movements | Baseline, 6 months
  The Choice Reaction Time subtest from the CANTAB assessment will be used to measure motor changes and bradykinesia.
Changes in cognitive ability | Baseline
  Cognitive ability will be measured using the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV).

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Napoli E, Flores A, Mansuri Y, Hagerman RJ, Giulivi C. Sulforaphane improves mitochondrial metabolism in fibroblasts from patients with fragile X-associated tremor and ataxia syndrome. Neurobiol Dis. 2021 Sep;157:105427. doi: 10.1016/j.nbd.2021.105427. Epub 2021 Jun 19. PMID 34153466
- [Background] Uddin MS, Mamun AA, Jakaria M, Thangapandiyan S, Ahmad J, Rahman MA, Mathew B, Abdel-Daim MM, Aleya L. Emerging promise of sulforaphane-mediated Nrf2 signaling cascade against neurological disorders. Sci Total Environ. 2020 Mar 10;707:135624. doi: 10.1016/j.scitotenv.2019.135624. Epub 2019 Nov 21. PMID 31784171
- [Background] Berry-Kravis EM, Harnett MD, Reines SA, Reese MA, Ethridge LE, Outterson AH, Michalak C, Furman J, Gurney ME. Inhibition of phosphodiesterase-4D in adults with fragile X syndrome: a randomized, placebo-controlled, phase 2 clinical trial. Nat Med. 2021 May;27(5):862-870. doi: 10.1038/s41591-021-01321-w. Epub 2021 Apr 29. PMID 33927413

DOCUMENTS (1):
  • Informed Consent Form (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT05233579/ICF_000.pdf